CLINICAL TRIAL: NCT06193837
Title: Prophylactic Antibiotic in Non-complicated Low Risk Laparoscopic Cholecystectomy; Is it Worthy? A Prospective Randomized Comparative Study.
Brief Title: Prophylactic Antibiotic in Non-complicated Low Risk Lap Cholecystectomy (LC)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Mohammed Ali, Assiut Lecturer, Assiut University
Other Study IDs: Prophylactic Antibiotic in LC
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: Antibiotic; Lap cholecystectomy
MeSH Terms: interventions — Amoxicillin-Potassium Clavulanate Combination; Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Having prophylactic antibiotic in laparoscopic cholecystectomy
  Interventions: Drug: Augmentin
- Group 2: Not having prophylactic antibiotics in laparoscopic cholecystectomy

INTERVENTIONS:
Drug: Augmentin — Use of prophylactic antibiotics in lap cholecystectomy
  Other Names: laparoscopy
  Groups: Group 1

SUMMARY:
To Compare between outcomes of Antibiotic Prophylaxis and No antibiotic prophylaxis in non-complicated low risk laparoscopic cholecystectomy

DETAILED DESCRIPTION:
There is no doubt that Laparoscopic cholecystectomy (LC) is the surgery of choice in cholelithiasis [1].

Routine antibiotic prophylaxis in LC decreases the rate of intra and post operative infections specifically the Surgical site infection (SSI) [2]. However, the rate of antibiotic side effects remains considerable, mainly antibiotic resistance to the commonly used antibiotics as Cefoperazone and other antibiotics used in routine prophylaxis [3]. So Some studies proved that No need for antibiotic prophylaxis [4]. In spite, no antibiotic prophylaxis may lead to infections mainly SSI and prolongation of hospitalization time [5]. However None of these studies has proved Superiority over the other and stills a matter of controversy [6]. For this reason more efforts are directed to limit the use of antibiotic in non complicated low risk laparoscopic cholecystectomy. Prophylaxis in this study is directed to start from time of admission till 1 month post operative. In our study we Follow both outcomes to compare between both techniques

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female at the Age of 18 years or above.
* Symptomatic gall bladder stones.
* Ultrasonography shows gall bladder stones.
* Uncomplicated chronic calculous cholecystitis

Exclusion Criteria:

* Complicated gall bladder stones.
* Malignant gall bladder mass
* Laparoscopic cholecystectomy with Common Bile Duct (CBD) exploration.
* Absolute contraindications to LC like cardiovascular, pulmonary disease, coagulopathies and end stage liver disease.
* The cases of Laparoscopic Cholecystectomy conversion to Open Cholecystectomy due to equipment failure.
* Immunocompromised patients as Uncontrolled DM, HIV and patients on certain medications as corticosteroids and chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients with symptomatic chronic calcular cholecystitis with age above 18 years and fit for surgery. They should be with low-risk (Not immuno-compromized) and non-complicated cases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare between infection rate at both groups | Baseline
  Group 1; Prophylactic Antibiotics in LC and Group 2; No prophylactic antibiotics in LC
Hospitalization time | Baseline
  Group 1; Prophylactic Antibiotics in LC and Group 2; No prophylactic antibiotics in LC

SECONDARY OUTCOMES:
Improve quality of life to reduce mortality and morbidity in patients with chronic cholecystitis | Baseline
  Group 1; Prophylactic Antibiotics in LC and Group 2; No prophylactic antibiotics in LC

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M. Mohammad Sayed, Dr, Study Director — General Surgery department of Assiut University; Ahmed M. Ibrahim Taha, Dr, Study Director — General Surgery department of Assiut University

REFERENCES:
- [Background] Kim HJ, Kang SH, Roh YH, Kim MC, Kim KW. Are prophylactic antibiotics necessary in elective laparoscopic cholecystectomy, regardless of patient risk? Ann Surg Treat Res. 2017 Aug;93(2):76-81. doi: 10.4174/astr.2017.93.2.76. Epub 2017 Jul 28. PMID 28835883
- [Background] Yan RC, Shen SQ, Chen ZB, Lin FS, Riley J. The role of prophylactic antibiotics in laparoscopic cholecystectomy in preventing postoperative infection: a meta-analysis. J Laparoendosc Adv Surg Tech A. 2011 May;21(4):301-6. doi: 10.1089/lap.2010.0436. Epub 2011 Mar 28. PMID 21443433